CLINICAL TRIAL: NCT06779929
Title: Comparative Study of Tirzepatide vs Dulaglutide (SURPASS CVOT) or Semaglutide on Major Cardiovascular Events in Participants With Type 2 Diabetes
Brief Title: Comparative Study of Tirzepatide Versus Dulaglutide (SURPASS CVOT) or Semaglutide on Major Cardiovascular Events in Participants With Type 2 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elisabetta Patorno, MD, DrPH, Brigham and Women's Hospital
Other Study IDs: 2024P001317
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Tirzepatide; Dulaglutide; Type 2 diabetes; Cardiovascular disease; Myocardial infarction; Stroke; Mortality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Myocardial Infarction; Stroke | interventions — Tirzepatide; dulaglutide; semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tirzepatide: Patients who initiated tirzepatide with no use in the prior 180 days
  Interventions: Drug: Tirzepatide
- Dulaglutide: Patients who initiate dulaglutide with no use in the prior 180 days
  Interventions: Drug: Dulaglutide
- Semaglutide: Patients who initiate semaglutide with no use in the prior 180 days
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide
  Groups: Tirzepatide
Drug: Dulaglutide — Dulaglutide
  Groups: Dulaglutide
Drug: Semaglutide — Semaglutide
  Groups: Semaglutide

SUMMARY:
This cohort study was initiated to emulate the design of the SURPASS-CVOT trial using observational analogues of the trial design components in a study based on insurance claims data.

DETAILED DESCRIPTION:
Recent evidence suggests that the metabolic effects of glucagon-like peptide-1 receptor agonists (GLP-1RA) can be enhanced by combining them with the actions of other entero-pancreatic hormones, such as glucose-dependent insulinotropic polypeptide (GIP) and/or glucagon. Tirzepatide is a once-weekly GIP/GLP-1RA, approved for the treatment of type 2 diabetes in May 2022.

The Study of Tirzepatide Compared With Dulaglutide on Major Cardiovascular Events in Participants With Type 2 Diabetes (SURPASS-CVOT; NCT04255433) is an event-driven, randomized, double- blind, active comparator, parallel-group study, to evaluate cardiovascular (CV) outcomes with tirzepatide treatment in people with type 2 diabetes (T2D) and established atherosclerotic CV disease (ASCVD) compared with dulaglutide treatment, stratified by baseline sodium-glucose cotransporter-2 (SGLT2) inhibitors use. SURPASS-CVOT was designed to establish CV protection with tirzepatide by demonstrating noninferiority of tirzepatide to dulaglutide, and also to determine whether tirzepatide produces a greater CV benefit than dulaglutide (superiority analysis).

This new user active comparator cohort study aims to emulate the SURPASS-CVOT trial using insurance claims data. Trial design parameters were adapted in claims data using observational analogues for eligibility criteria, treatment strategies, treatment assignment, follow-up start, follow-up end, outcome, and causal contrast. We also conducted HbA1c-adjusted analyses among those with HbA1c values (54% of population).

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2D who were new users of tirzepatide or new users of dulaglutide
* AND established ASCVD defined as:

  * History of Myocardial Infarction (MI) or MI sequela
  * Unstable or stable angina
  * Coronary atherosclerosis disease or procedures
  * Ischemic stroke
  * Peripheral arterial disease or procedures
  * Atherosclerotic cerebrovascular disease or cerebrovascular procedures
  * Lower-limb amputation
* Age >= 40 years old
* Patients with at least 180 days of continuous health plan enrollment before and including the treatment initiation date

Exclusion Criteria:

* Patients with Type 1 diabetes mellitus
* Patients with missing age or sex information
* Patients with history of proliferative diabetic retinopathy, panretinal photocoagulation, vitreous hemorrhage, or intravitreal anti-VEGF injection
* Patient within history of left ventricular assisted device (LVAD) or heart transplant
* Patients with any previous organ transplants
* Patients with acute of chronic pancreatitis
* Patients with gastroparesis, bowel obstruction or bariatric surgery
* Patient with CKD Stage 5, end stage kidney disease, kidney transplant, or hemodialysis
* Patients with multiple endocrine neoplasm syndrome type 2 (MEN-2)
* Patient with cancer
* Pregnant women
* Patient with diabetic ketoacidosis or HONK within the last year to treatment initiation
* Patients with acute hepatitis within the last year to treatment initiation
* Patients with elevated serum calcitonin level within the last year to treatment initiation
* Previous exposure to GLP-1RA or pramlintide during the 180-days washout period and including treatment initiation date
* Patients with severe hypoglycemia within the last 6 months to treatment initiation
* Patients with hospitalization for heart failure within the last 60 days to treatment initiation
* Patient with acute coronary syndrome, ischemic stroke, peripheral arterial disease, or coronary or cerebrovascular procedure within the last 60 days to treatment initiation
* Patients with prescription dispensing for both tirzepatide and dulaglutide on treatment initiation date

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients > 40 years old with T2D and established atherosclerotic cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite CV outcome | From treatment initiation to end of follow up, up to 48 months.
  Composite CV outcome includes myocardial infarction, stroke, and all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Nicholls SJ, Bhatt DL, Buse JB, Prato SD, Kahn SE, Lincoff AM, McGuire DK, Nauck MA, Nissen SE, Sattar N, Zinman B, Zoungas S, Basile J, Bartee A, Miller D, Nishiyama H, Pavo I, Weerakkody G, Wiese RJ, D'Alessio D; SURPASS-CVOT investigators. Comparison of tirzepatide and dulaglutide on major adverse cardiovascular events in participants with type 2 diabetes and atherosclerotic cardiovascular disease: SURPASS-CVOT design and baseline characteristics. Am Heart J. 2024 Jan;267:1-11. doi: 10.1016/j.ahj.2023.09.007. Epub 2023 Sep 25. PMID 37758044